CLINICAL TRIAL: NCT02098174
Title: Pharmacokinetics of MP-3180 in Healthy Volunteers
Acronym: Pilot 1A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ORFM-1A
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Glomerular Filtration Rate; Acute Kidney Injury
Keywords: Glomerular Filtration Rate; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy participants (Experimental): MP-3180 (1 µmol/kg or 0.372 mg/kg) was administered by IV injection (2.5 mL to 3.5 mL for participant weights of 70 kg to 91 kg) over 2 minutes, followed by a 10 mL saline flush IV over 2 minutes. The iohexol comparator (Omnipaque 300, 5 mL) was then administered by IV injection over 2 minutes, followed by a 10 mL saline flush IV over 2 minutes.
  Interventions: Drug: MP-3180; Other: Iohexol comparator

INTERVENTIONS:
Drug: MP-3180 — MP-3180 (1 µmol/kg or 0.372 mg/kg) (fluorescent tracer agent) was administered by IV injection (2.5 mL to 3.5 mL for participant weights of 70 kg to 91 kg) over 2 minutes, followed by a 10 mL saline flush IV over 2 minutes.
Other: Iohexol comparator — Iohexol (Omnipaque 300, 5 mL) was administered by IV injection over 2 minutes, followed by a 10 mL saline flush IV over 2 minutes.

SUMMARY:
The purpose of this study was to investigate the pharmacokinetics of MP-3180 (1 µmol/kg) compared to the pharmacokinetics of iohexol (5 mL of a 300 mg iodine (I)/mL solution) in healthy adult participants. The secondary objective was to evaluate the safety and tolerability of MP-3180 in healthy adult participants.

DETAILED DESCRIPTION:
Single-dose pharmacokinetics were characterized in sixteen (16) healthy, adult male participants in this Phase 1, open-label study following the administration of a single, intravenous 1 µmol/kg dose over 2 minutes followed by 10 mL saline under fasting conditions. Iohexol (Omnipaque-300, 5 mL of a 300 mg I/mL solution) was also administered over 2 minutes followed by 10 mL of saline. The pharmacokinetics of MP-3180 and iohexol was assessed by statistical comparison of pharmacokinetic parameters derived from plasma concentration-time curves and urine recovery data.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 22 years of age or older
* 2. Sex: males and not of childbearing potential females
* 3. Capable of informed consent
* 4. Weight restrictions:

  * a. at least 50 kg (110 lbs) for men
  * b. at least 48 kg (106 lbs) for women
  * c. All participants will have a Body Mass Index (BMI) less than or equal to 33 but greater than or equal to 19
* 5. All participants should be judged by the Principal Investigator or Medical Sub-Investigator physician as normal and healthy during a pre-study medical evaluation performed within 28 days of the initial dose of study medication

Exclusion Criteria:

* 1. Institutionalized participants will not be used
* 2. Social habits:

  * a. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
  * b. Ingestion of any vitamins or herbal supplement within 7 day prior to the initial dose of study medication.
  * c. Any significant change in dietary or exercise habits within the 48 hours prior to the initial dose of study medication.
  * d. History of drug and/or alcohol abuse within the past year, unless currently enrolled in an abstinence program.
* 3. Use of any prescription or over-the-counter (OTC) medications within the 7 days prior to the initial dose of study medication.
* 4. History of any significant cardiovascular disease, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic (including any history of seizure disorder), psychological, musculoskeletal disease or malignancies unless deemed not clinically significant by the Principal Investigator or Medical Sub-Investigator.
* 5. Acute illness at the time of either the pre-study medical evaluation or dosing.
* 6. Not within normal limits or clinically significant for lab testing
* 7. Any reason which, in the opinion of the Principal Investigator or Medical Sub-Investigator, would prevent the participant from safely participating in the study.
* 8. Donation or loss of blood or plasma: 50 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication.
* 9. Intolerance to venipuncture.
* 10. Participants who have received an investigational drug within 30 days prior to the initial dose of study medication.
* 11. History of allergy or hypersensitivity to MP-3180 or iohexol, or other related products, or any of the inactive ingredients.
* 12. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Principal Investigator or Medical Sub-Investigator, could contraindicate the participant's participation in this study.
* 13. History of allergy or hypersensitivity to iodine containing contrast media or drugs.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Total plasma clearance of MP-3180 and iohexol | Pre-dose and the following times after dosing: 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. Total plasma clearance (the volume of plasma cleared of the drug over time) was calculated as: Clp = Dose/ AUC∞.
Renal clearance of MP-3180 and iohexol | Pre-dose and each time the participant voided up to 720 minutes post dose
  Urine samples were collected pre-dose (time 0) and 5 mL urine samples were collected each time the subject voided. The total volume of urine excreted was recorded until 12 hours post-dose, and analyzed using validated analytical methods. Renal clearance (the volume of plasma cleared of the drug by the kidneys over time) was calculated as: CLr = Ae/ AUClast, where Ae is the cumulative amount of analyte excreted in urine over the sampling interval.
Maximum Plasma Concentration (Cmax) for MP-3180 and iohexol | Pre-dose and the following times after dosing: 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. Maximum plasma concentration (Cmax; measured in ng/mL) was directly determined from the concentration-time data.
Time to Maximum Plasma Concentration (Tmax) for MP-3180 and iohexol | Pre-dose and the following times after dosing: 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The time to maximum plasma concentration (Tmax; measured in hours) was directly determined from the concentration-time data.
The terminal rate constant for MP-3180 and iohexol | Pre-dose and the following times after dosing: 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The terminal rate constant (λz) was determined by linear regression of the terminal linear phase of the log plasma concentration-time profile.
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration for MP-3180 and iohexol | Pre-dose and the following times after dosing: 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The area under the plasma concentration-time curve (ng*hr/mL) was estimated from time 0 to the last measurable concentration using noncompartmental analyses.
Area under the plasma concentration-time curve from time zero to infinity for MP-3180 and iohexol | Pre-dose and the following times after dosing: 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The area under the plasma concentration-time curve (ng*hr/mL) from time 0 to infinity was calculated as: AUC∞ = AUClast + LQC/λz where LQC is the predicted concentration (based on the terminal regression) at the time of the last measurable concentration.
The elimination half-life of MP-3180 and iohexol | Pre-dose and the following times after dosing: 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The elimination half-life (the time required for the concentration of the drug to reach half of its original value) was calculated as t1/2 λz= ln(2)/ λz.

SECONDARY OUTCOMES:
Incidence of adverse events | 1, 3, and 8 hours after dosing, and within 2 weeks after the final study dose
  An adverse event (AE) was defined as any untoward medical occurrence in a study subject after study drug administration and that did not necessarily have a causal relationship with this treatment.
Number of laboratory values that fall outside of pre-specified normal ranges | Pre-dose and within 2 weeks after the final study dose
  Blood samples were collected and analyzed for hematology and clinical chemistry. Out of range values were documented.

OTHER OUTCOMES:
Correlation between the plasma clearance of MP-3180 and the plasma clearance of iohexol | Pre-dose and 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. Mean concentrations over time were determined.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dowling, Ph.D., Principal Investigator — University of Maryland; Richard B. Dorshow, Ph.D., Study Director — MediBeacon, LLC
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No